CLINICAL TRIAL: NCT01125852
Title: Supplementary Angiographic Embolization for Peptic Ulcer Bleeding: A Randomized Controlled Trial
Brief Title: Supplementary Angiographic Embolization for Peptic Ulcer Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Stig Borbjerg Laursen, MD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-20090086
Record Dates: First submitted 2010-05-10; First posted 2010-05-19 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Peptic Ulcer Hemorrhage
Keywords: Peptic ulcer hemorrhage; Peptic ulcer bleeding; Angiographic embolization; Arterial embolization; Angiography
MeSH Terms: conditions — Peptic Ulcer Hemorrhage | interventions — Embolization, Therapeutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Active Comparator): Patients in this group are treated with usual therapeutic endoscopy including endoscopic combination therapy and 72 hours intravenous proton pump inhibitor. Within 24 hours from the therapeutic endoscopy they receive supplementary angiographic embolization.
  Interventions: Procedure: Angiographic embolization
- Control group (Active Comparator): Patients in this arm receive standard treatment including therapeutic endoscopy with endoscopic combination therapy followed by 72 hours intravenous proton pump inhibitor.
  Interventions: Procedure: Therapeutic endoscopy

INTERVENTIONS:
Procedure: Angiographic embolization — Patients in the intervention arm receive supplementary angiographic embolization within 24 hours from the therapeutic endoscopy.
  Other Names: Therapeutic angiography; Arterial embolization; Transcatheter arterial embolization; Embolization
  Arms: Intervention group
Procedure: Therapeutic endoscopy — Patients are treated with standard therapeutic upper endoscopy including endoscopic combination therapy.
  Arms: Control group

SUMMARY:
Peptic ulcer bleeding is a common disorder. Despite optimal endoscopic and medical treatment, there is a high risk of rebleeding and high mortality. In this study the investigators examine whether combined endoscopic haemostasis and angiographic embolization resolves in a better outcome than the traditional use of endoscopic haemostasis alone. The study is a randomised controlled trail.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs of upper GI-bleeding
* Endoscopic verified high-risk ulcer (Forrest I-IIb)
* Primary haemostasis achieved

Exclusion Criteria:

* Expected lifetime < 1 month
* Upper GI-cancer found at endoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2009-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Composite Endpoint | Meassured after a week from primary therapeutic endoscopy
  Patients are classified into groups depending on the worst outcome:
  1. No clinical signs of rebleeding and requirement of two or less blood transfusions after circulatory stabilization and obtained hemoglobin > 5,9mmol/L.
  2. No clinical signs of rebleeding and requirement of more than two blood transfusions after circulatory stabilization and obtained hemoglobin > 5,9mmol/L.
  3. Rebleeding and achieved secondary haemostasis by endoscopy or angiographic embolization.
  4. Rebleeding requiring surgery.
  5. Patients who have died.
  Results are compared using the Wilcoxon rank sum test.

SECONDARY OUTCOMES:
Mortality | 1 month
  Patients who have died within af month from therapeutic endoscopy.
Rebleeding | 1 month
  Rebleeding from ulcer confirmed by endoscopy, angiography or surgery within a month from therapeutic endoscopy.
Blood transfusion | 1 month
  Amount of received blood transfusions after circulatory stabilization and obtained hemoglobin > 5,9mmol/L. Patients will only receive blood transfusion if hemoglobin < 6,0mmol/L
Surgical haemostasis | 1 month
  Rebleeding requiring surgical haemostasis within a month from therapeutic endoscopy.
Endoscopic/other haemostatic retreatment | 1 month
  Rebleeding confirmed by endoscopy or angiography and achieved secondary haemostasis by endoscopy or angiographic embolization.
Duration of hospitalization | Estimated 4 days
  Time from hospitalization to discharge.
Thromboembolic complications | 1 month
  Occurence of thromboembolic complications due to angiographic embolization, surgery or therapeutic endoscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Laursen SB, Hansen JM, Andersen PE, Schaffalitzky de Muckadell OB. Supplementary arteriel embolization an option in high-risk ulcer bleeding--a randomized study. Scand J Gastroenterol. 2014 Jan;49(1):75-83. doi: 10.3109/00365521.2013.854829. Epub 2013 Nov 21. PMID 24256098